CLINICAL TRIAL: NCT05709834
Title: Effects of Autogenic Training on Blood Pressure and Anxiety in Females With Pre-eclampsia
Brief Title: Autogenic Training Effects on Pre-eclampsia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Adeela
Record Dates: First submitted 2023-01-04; First posted 2023-02-02 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Pre-Eclampsia
MeSH Terms: conditions — Pre-Eclampsia | interventions — Autogenic Training; Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Autogenic training (Experimental): It consists of patients who will receive autogenic training and conventional treatment with the frequency of 3 times per week for 4 weeks.
  Interventions: Other: Autogenic training
- Control group (Other): Its consists of patients who will receive conventional treatment with the frequency of 3 sessions per week
  Interventions: Other: Conventional treatment

INTERVENTIONS:
Other: Autogenic training — Relaxation procedures will be performed in the following steps: First step - preparation: Each pre-eclamptic woman will be instructed about this method of treatment and its importance for reducing blood pressure to gain her confidence and cooperation during treatment. Second step - AT: The session began with a few minutes of mental relaxation as the patient will be asked to imagine herself in a lovely place that makes her relaxed. Each session include 18 exercises combining both relaxation and auto-suggestion (limb heaviness exercise, limb warmth exercise, cardiac exercise, respiration exercise, solar plexus warmth exercise, and "forehead cooling" exercise).
  About 30 sec will be allowed for each exercise and a further 30-40 sec will allowed for continuing attention focusing by the patient. Third step - termination
  Arms: Autogenic training
Other: Conventional treatment — Patients will receive conventional treatment
  Other Names: Control group
  Arms: Control group

SUMMARY:
The purpose of study is to find the effects of autogenic training on blood pressure and anxiety in preeclampsia females. There is little of evidence to allow conclusions about effectiveness of autogenic training on preeclampsia Therefore this study will add to the growing body of knowledge that if autogenic training is better than any other protocol for preeclampsia and anxiety then it should be a choice of therapy treatment. This study can provide help pregnant females and other society members to think about treatment of preeclampsia and anxiety other than medical approach.

DETAILED DESCRIPTION:
Pre-eclampsia is a disorder of pregnancy characterized by the onset of high blood pressure and often a significant amount of protein in the urine. When it arises, the condition mostly begins after 20 weeks of pregnancy. In severe cases of the disease there may be red blood cell breakdown, a low blood platelet count, impaired liver function, kidney dysfunction, swelling, shortness of breath due to fluid in the lungs, or visual disturbances. Pre-eclampsia increases the risk of undesirable outcomes for both the mother and the fetus. Pre-eclampsia affects approximately 2-8% of all pregnancies worldwide. Pre-eclampsia is much more common in women who are pregnant for the first time or have obesity, diabetes and autoimmune disease.

Randomized controlled trial (RCT) will be conducted to find the effects of autogenic training on blood pressure and anxiety in females having pre-eclampsia, the data will be collected from National Hospital and Sofia clinic via sphygmomanometer and DASS-21 scale. Sample size of 26 females is taken. Non probability convenient sampling will be used. A written consent form will be taken from participants meeting inclusion criteria and will be randomly allocated into two groups through lo1.ttery method to either Group A or Group B. Treatment will be given 3 times per week for 4 weeks. Sphygmomanometer will be used to check the blood pressure reading and DASS-21 questionnaire will be used to access anxiety in the females. All participants in both groups will be evaluated before and after the treatment program. Total duration of the study will be ten months. Data will be analyzed by using SPSS 21.

ELIGIBILITY:
Inclusion Criteria:

* Diagnose Women with pre-eclampsia
* Blood pressure value more than 90/140
* 2nd trimester
* Age of 25 to 35 years

Exclusion Criteria:

* Women with cardiorespiratory diseases and diabetes
* Previous history of preterm labor or abortion
* History of serious mental illness

Ages: 25 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 26 (Actual)
Dates: Start 2022-01-15 (Actual); Primary Completion 2023-02-25 (Actual); Study Completion 2023-03-15 (Actual)

PRIMARY OUTCOMES:
Blood Pressure | 4th week
  The sphygmomanometer is an objective tool used to measure the blood pressure.it consist of the inflatable rubber cuff, which is wrapped around the upper arm connected to an appratus that records pressure. The sounds are detected by the doctor using a stethoscope.it is also called blood pressure gauge The validity or specificity of sphygnomanometer is 0.7.
Anxiety | 4th week
  The Depression Anxiety Stress Scales (DASS-21) was designed to measure the core symptoms of depression, anxiety and stress and has demonstrated excellent psychometric properties across studies. Each of the three DASS-21 scales contains 7 items, divided into subscales with similar content. The depression scale assesses dysphoria, hopelessness and lack of interest. The anxiety scale assesses autonomic arousal, skeletal muscle effects and situational anxiety and the stress scale assesses difficulty relaxing, agitated, and impatient. The validity of scale is 0.90.

CONTACTS AND LOCATIONS:
Overall Officials: Adeela Arif, Mphil, Principal Investigator — Riphah International University
Locations (1):
- Riphah International university, Lahore, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Awad MA, Hasanin ME, Taha MM, Gabr AA. Effect of stretching exercises versus autogenic training on preeclampsia. J Exerc Rehabil. 2019 Feb 25;15(1):109-113. doi: 10.12965/jer.1836524.262. eCollection 2019 Feb. PMID 30899745
- [Background] Lu HQ, Hu R. The role of immunity in the pathogenesis and development of pre-eclampsia. Scand J Immunol. 2019 Nov;90(5):e12756. doi: 10.1111/sji.12756. Epub 2019 Sep 9. PMID 30739345
- [Background] Soto-Balbuena C, Rodriguez MF, Escudero Gomis AI, Ferrer Barriendos FJ, Le HN, Pmb-Huca G. Incidence, prevalence and risk factors related to anxiety symptoms during pregnancy. Psicothema. 2018 Aug;30(3):257-263. doi: 10.7334/psicothema2017.379. PMID 30009746
- [Background] Abedian Z, Soltani N, Mokhber N, Esmaily H. Depression and anxiety in pregnancy and postpartum in women with mild and severe preeclampsia. Iran J Nurs Midwifery Res. 2015 Jul-Aug;20(4):454-9. doi: 10.4103/1735-9066.161013. PMID 26257800
- [Background] Horsley KJ, Tomfohr-Madsen LM, Ditto B, Tough SC. Hypertensive Disorders of Pregnancy and Symptoms of Depression and Anxiety as Related to Gestational Age at Birth: Findings From the All Our Families Study. Psychosom Med. 2019 Jun;81(5):458-463. doi: 10.1097/PSY.0000000000000695. PMID 30985405